CLINICAL TRIAL: NCT05891158
Title: An Open-Label, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, Tolerability, and Pharmacodynamics in Response to a Single Subcutaneous Dose of Fazirsiran (TAK-999) in Subjects With or Without Hepatic Impairment
Brief Title: A Study About Fazirsiran in People With and Without Liver Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-999-1001; 2023-503735-17-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1, Mild HI: Fazirsiran 200 mg (Experimental): Participants with mild hepatic impairment (HI) will receive fazirsiran 200 milligrams (mg) subcutaneous (SC) injection on Day 1.
  Interventions: Drug: Fazirsiran
- Arm 2, Moderate HI: Fazirsiran 200 mg (Experimental): Participants with moderate HI will receive fazirsiran 200 mg SC injection on Day 1. The dose may be modified after review of available safety and PK data by the sponsor study team in consultation with the investigator.
  Interventions: Drug: Fazirsiran
- Arm 3, Severe HI: Fazirsiran 200 mg (Experimental): Participants with severe HI will receive fazirsiran 200 mg SC injection on Day 1. The dose may be modified after review of available safety and PK data by the sponsor study team in consultation with the investigator.
  Interventions: Drug: Fazirsiran
- Arm 4, Normal Hepatic Function: Fazirsiran 200 mg (Experimental): Participants with normal hepatic function will receive fazirsiran 200 mg SC injection on Day 1. The dose may be modified after review of available safety and PK data by the sponsor study team in consultation with the investigator.
  Interventions: Drug: Fazirsiran

INTERVENTIONS:
Drug: Fazirsiran — Fazirsiran SC injection
  Other Names: TAK-999

SUMMARY:
The main aim of this study is to learn how the body processes fazirsiran (pharmacokinetics [PK]) in people with mild, moderate, or severe liver problems, compared to people with normal liver function.

The study will include participants with liver scarring (cirrhosis) and mild, moderate, or severe liver problems, and participants with normal liver function. All participants will be given 1 injection of fazirsiran and will be followed up for 6 months after the fazirsiran injection.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria for All Participants

* A 12-lead ECG at screening that, in the opinion of the investigator, has no abnormalities that compromise the participant's safety in this study.
* No abnormal finding of clinical relevance at screening or before dosing that in the opinion of the investigator could adversely impact participant safety during the study or adversely impact study results.

Key Inclusion Criteria for Participants with Hepatic Impairment:

* The participant is 18 to 75 years of age inclusive at the time of signing the informed consent form (ICF).
* The participant has a body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 40.0 kilograms per square meter (kg/m^2) at screening.
* Aside from HI, the participant must be sufficiently healthy for study participation based upon medical history, physical examination, vital signs, electrocardiograms (ECGs), and screening clinical laboratory profiles, as deemed by the investigator or designee.
* Diagnosis of chronic (example, imaging, biopsy, etc.) stable hepatic insufficiency for at least 3 months before screening with features of cirrhosis due to any etiology according to medical history. HI must be stable, that is, no significant changes in hepatic function or clinical status in the 30 days preceding screening (or since the last visit if within 3 months before screening) and with treatment with stable doses of medication.
* Has a Child-Turcotte-Pugh (CTP) score confirmed by 2 tests as follows:
* Arm 1: Mild HI, CTP Class A: >=5 and <=6
* Arm 2: Moderate HI, CTP Class B: >=7 and <=9
* Arm 3: Severe HI, CTP Class C: >=10 and <=15
* It must be confirmed that the participant does not have hepatocellular carcinoma (HCC).

Key Inclusion Criterion for Participants with Mild Hepatic Impairment • The participant has pulmonary status meeting criteria of percent predicted forced expiratory volume in the first second of expiration (ppFEV1) >=80 percent and percent predicted diffusing capacity of the lungs for carbon monoxide adjusted for hemoglobin (ppDLCOhgb) >=75%, based on pulmonary function test (PFT) at screening conducted as per American Thoracic Society (ATS)-European Respiratory Society (ERS) criteria.

Key Inclusion Criterion for Participants with Moderate and Severe Hepatic Impairment

• The participant has pulmonary status meeting the criteria defined in the protocol based on PFT at screening conducted as per ATS-ERS criteria.

Key Inclusion Criteria for Participants with Normal Hepatic Function

* The participant is 18 to 85 years of age inclusive, at the time of signing the ICF.
* The participant has a BMI >=18.0 and <=40.0 kg/m^2, at screening. Participants will be matched to participants with HI by BMI (±15%).
* AAT level at or above the lower end of the reference range (above or equal to 16.6 micromole (mcM) or 90 milligram per deciliter [mg/dL]) at screening.
* The participant has normal liver tests including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and total bilirubin (TBILI) <=1.2 x upper limit of the normal range (ULN) at screening and check-in.
* The participant has pulmonary status meeting criteria of ppFEV1 >=80%, and ppDLCOhgb >=75%, based on PFT at screening conducted as per ATS- ERS criteria.

Exclusion Criteria:

Key Exclusion Criteria for All Participants:

* The participant has uncontrolled hypertension (systolic blood pressure [BP] >170 mm Hg and diastolic BP >100 millimeter of mercury [mmHg] at screening). Participants may be rescreened once BP is successfully controlled.
* The participant has a history of torsades de pointes, ventricular rhythm disturbances (example, ventricular tachycardia or fibrillation), heart block (excluding first-degree block, being pulse rate [PR] interval prolongation only), congenital long QT syndrome or new ST segment elevation or depression or new Q wave on ECG. Participants with a history of atrial arrhythmias should be discussed with the medical monitor.
* The participant has symptomatic heart failure (per New York Heart Association guidelines) or severe heart failure with reduced ejection fraction (EF <20%), unstable angina, myocardial infarction, transient ischemic attack, or cerebrovascular accident within 6 months before screening.
* The participant is expected to have severe and unavoidable high-level exposure to inhaled pulmonary toxins during the study.
* The participant has had a recent lower respiratory tract infection, such as pneumonia, within the last 6 months before screening.
* The participant has a history of malignancy within the last 1 year, except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer. Participants with other curatively treated malignancies who have no evidence of metastatic disease and have been disease-free for >1 year may enter the study after approval by the medical monitor.
* The participant has a history of thromboembolic disease (including deep vein thrombosis or pulmonary embolism) within 6 months of screening.

Key Exclusion Criteria for Participants with Hepatic Impairment:

* The participant has a history of gastric or esophageal variceal bleeding within the past 6 months of dosing and for which varices have not been adequately treated with medication and/or endoscopic procedures.
* The participant has grade >2 hepatic encephalopathy assessed using the West Haven criteria.
* The participant has evidence of hepatopulmonary syndrome or portal-pulmonary hypertension.
* The participant has portal vein thrombosis, transjugular intrahepatic portosystemic shunt (TIPS), or surgical portosystemic shunt.
* The participant has required endoscopic treatment of esophageal or gastric varices or paracentesis to control ascites within the last 3 months of dosing.
* The participant has chronic hepatitis B (hepatitis B surface antigen positive, or positive for both hepatitis B surface antibody and hepatitis B core antibody but negative for hepatitis B surface antigen); or has chronic or incompletely or unsuccessfully treated hepatitis C (as demonstrated by a positive hepatitis C antibody and positive polymerase chain reaction [PCR]).
* The participant has any of the following clinically significant abnormal parameters at screening:

  * ALT or AST levels >250 units per liter (U/L) at screening.
  * Estimated glomerular filtration rate <45 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for Fazirsiran | From pre-dose up to Month 6 post-dose
Area Under the Plasma Concentration-time Curve from Time 0 to Infinity (AUC0-inf) for Fazirsiran | From pre-dose up to Month 6 post-dose
Maximum Observed Plasma Concentration (Cmax) for Fazirsiran | From pre-dose up to Month 6 post-dose

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From the first dose of study drug up to end of follow-up (up to 6 months)
Number of Participants With Clinically Significant Abnormal Values for Laboratory Parameters | From the first dose of study drug up to end of follow-up (up to 6 months)
Number of Participants With Clinically Significant Abnormal Values for Vital Signs Parameters | From the first dose of study drug up to end of follow-up (up to 6 months)
Number of Participants With Clinically Significant Abnormal Values for Electrocardiogram (ECG) Parameters | From the first dose of study drug up to end of follow-up (up to 6 months)
Number of Participants With Clinically Significant Abnormal Values for Pulmonary Function Parameters | From the first dose of study drug up to end of follow-up (up to 6 months)
Number of Participants With Injection Site Reaction | From the first dose of study drug up to end of follow-up (up to 6 months)
Amount of Drug Excreted in Urine From Time 0 to Time 24 hours (Ae0-24hrs) for Fazirsiran | Pre-dose, 0 to 24 hours post-dose
Amount of Drug Excreted in Urine From Time 0 to Time 6 hours (Ae0-6hrs) for Fazirsiran | Pre-dose, 0 to 6 hours post-dose
Amount of Drug Excreted in Urine From Time 6 to Time 24 hours (Ae6-24h) for Fazirsiran | From 6 to 24 hours post-dose
Percent of Recovered Drug in Urine Compared With the Dose (%Dose [u]) | Pre-dose, 0 to 24 hours post-dose
Renal Clearance (CLr) for Fazirsiran | Pre-dose, 0 to 24 hours post-dose
Absolute Change in Serum Alpha-1 Antitrypsin (AAT) at Nadir | From Day 1 Pre-dose Baseline up to end of follow-up (up to 6 months)
Percentage Change in Serum AAT at Nadir | From Day 1 Pre-dose Baseline up to end of follow up (up to 6 months)
Absolute Change in Serum AAT | From Day 1 Pre-dose Baseline and at Days 15, 29, 57
Percentage Change in Serum AAT | From Day 1 Pre-dose Baseline and at Days 15, 29, 57

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- CRU Hungary Kft, Kistarcsa, Hungary
- Slovakia (3):
  - Summit Clinical Research s.r.o., Bratislava
  - Summit Clinical Research s.r.o., Malacky
  - Summit Clinical Research s.r.o., Nové Zámky

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/3f603e5edec44979?idFilter=%5B%22TAK-999-1001%22%5D